CLINICAL TRIAL: NCT01081041
Title: A Randomized, Double-Blind, Phase 2 Safety Study of Cetuximab, Using ImClone Versus Boehringer Ingelheim Manufacturing Processes, in Combination With Cisplatin or Carboplatin and 5-Fluorouracil in the First-Line Treatment of Patients With Locoregionally Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Study in Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13611; I4E-MC-JXBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Safety Lead-In (cetuximab manufactured by ImClone) (Experimental): Cycle 1:
  Week 1 - Cetuximab 400 milligrams per square meter (mg/m^2) on Day 1; Cisplatin 100 mg/m^2 on Day 1 or carboplatin area under the curve (AUC) 5 on Day 1; 5-FU 1000 mg/m^2 on Days 1-4
  Week 2 - Cetuximab 250 mg/m^2 on Day 1
  Week 3 - Cetuximab 250 mg/m^2 on Day 1
  Cycle 2-6:
  Week 1 - Cetuximab 250 mg/m^2 on Day 1; Cisplatin 100 mg/m^2 on Day 1 or carboplatin AUC 5 on Day 1; 5-FU 1000 mg/m^2 on Days 1-4
  Week 2 - Cetuximab 250 mg/m^2 on Day 1
  Week 3 - Cetuximab 250 mg/m^2 on Day 1
  After 6 cycles, participants may then receive weekly cetuximab monotherapy 250 mg/m^2 until progression of disease, unacceptable toxicity, or another withdrawal criteria is met.
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-Fluorouracil
- Cetuximab manufactured by ImClone (Experimental): Cycle 1:
  Week 1 - Cetuximab 400 mg/m^2 on Day 1; Cisplatin 100 mg/m^2 on Day 1 or carboplatin AUC 5 on Day 1; 5-FU 1000 mg/m^2 on Days 1-4
  Week 2 - Cetuximab 250 mg/m^2 on Day 1
  Week 3 - Cetuximab 250 mg/m^2 on Day 1
  Cycle 2-6:
  Week 1 - Cetuximab 250 mg/m^2 on Day 1; Cisplatin 100 mg/m^2 on Day 1 or carboplatin AUC 5 on Day 1; 5-FU 1000 mg/m^2 on Days 1-4
  Week 2 - Cetuximab 250 mg/m^2 on Day 1
  Week 3 - Cetuximab 250 mg/m^2 on Day 1
  After 6 cycles, participants may then receive weekly cetuximab monotherapy 250 mg/m^2 until progression of disease, unacceptable toxicity, or another withdrawal criteria is met.
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-Fluorouracil
- Cetuximab manufactured by Boehringer Ingelheim (Experimental): Cycle 1:
  Week 1 - Cetuximab 400 mg/m^2 on Day 1; Cisplatin 100 mg/m^2 on Day 1 or carboplatin AUC 5 on Day 1; 5-FU 1000 mg/m^2 on Days 1-4
  Week 2 - Cetuximab 250 mg/m^2 on Day 1
  Week 3 - Cetuximab 250 mg/m^2 on Day 1
  Cycle 2-6:
  Week 1 - Cetuximab 250 mg/m^2 on Day 1; Cisplatin 100 mg/m^2 on Day 1 or carboplatin AUC 5 on Day 1; 5-FU 1000 mg/m^2 on Days 1-4
  Week 2 - Cetuximab 250 mg/m^2 on Day 1
  Week 3 - Cetuximab 250 mg/m^2 on Day 1
  After 6 cycles, participants may then receive weekly cetuximab monotherapy 250 mg/m^2 until progression of disease, unacceptable toxicity, or another withdrawal criteria is met.
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Cetuximab — Administered intravenously
  Other Names: Erbitux; LY2939777
Drug: Cisplatin — Administered intravenously
Drug: Carboplatin — Administered intravenously
Drug: 5-Fluorouracil — Administered intravenously
  Other Names: 5-FU

SUMMARY:
This study will begin with a 30 participant lead-in part: these 30 participants will receive cetuximab manufactured by ImClone on a weekly basis in combination with other chemotherapy drugs [cisplatin or carboplatin plus 5-fluorouracil (5-FU)] administered every 3 weeks. After 18 weeks, participants who benefit from this treatment may continue to receive cetuximab once-weekly until progression of the disease, an unacceptable side effect occurs, participants withdraw consent, or the study is closed.

In the second part of this study, 200 participants will be randomized in 2 arms:

* 100 participants will receive commercial cetuximab manufactured by ImClone (Group A)
* 100 participants will receive cetuximab manufactured by Boehringer Ingelheim (Group B).

All these 200 participants will receive other chemotherapy drugs (cisplatin or carboplatin plus 5-FU) administered every 3 weeks. After 18 weeks, participants who benefit from this treatment may continue to receive cetuximab once-weekly until progression of the disease, an unacceptable side effect occurs, participants withdraw consent, or the study is closed.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer that was confirmed by tissue biopsy or cytology
* Disease not suitable for local therapy
* Measurable or evaluable disease
* Karnofsky performance status (KPS) score of at least 70
* Organs are functioning well (bone marrow reserve, liver and kidney)
* Life expectancy of at least 12 weeks
* Signed informed consent document

Exclusion Criteria:

* Receiving another investigational medication within the last 30 days
* Prior chemotherapy, except if given as part of a multimodal treatment for locally advanced head and neck cancer that was completed more than 4 months prior to study entry.
* Nasopharyngeal carcinoma
* Previous treatment with monoclonal antibody therapy or other signal transduction inhibitors or epidermal growth factor receptor (EGFR) targeting therapy except for prior cetuximab treatment given as part of a multimodal treatment for locally advanced head and neck cancer that was completed more than 4 months prior to study entry.
* Uncontrolled high blood pressure
* Heart disease or had a heart attack within the last year
* Currently have an infection that requires for you to take an IV antibiotic
* Currently receiving other therapies for your cancer, such as chemotherapy, radiation therapy, immunotherapy, and hormonal therapy
* Medical or psychological condition that would not permit the participant to complete the study or sign informed consent
* Known drug abuse (with the exception of alcohol abuse)
* Known allergic reaction against any of the components of the study treatment
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment
* Have had another type of cancer within the last 2 years
* You are currently pregnant or breastfeeding
* You are considering becoming pregnant or fathering a child

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2010-06; Primary Completion 2013-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (26):
- United States (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fullerton, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Junction, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Weston, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Albany, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Abilene, Texas
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- Mexico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mérida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Soulieres D, Aguilar JL, Chen E, Misiukiewicz K, Ernst S, Lee HJ, Bryant K, He S, Obasaju CK, Chang SC, Chin S, Adkins D. Cetuximab plus platinum-based chemotherapy in head and neck squamous cell carcinoma: a randomized, double-blind safety study comparing cetuximab produced from two manufacturing processes using the EXTREME study regimen. BMC Cancer. 2016 Jan 14;16:19. doi: 10.1186/s12885-016-2064-0. PMID 26768732

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two-part study: Part 1 (single arm, safety lead-in) then Part 2 (parallel treatment comparison). All participants to complete 6 cycles of combination therapy then, if eligible, monotherapy. Participant flow presents those who completed study (died); those who were alive or death status unknown at data cut-off considered to not have completed study.
Groups:
- Part 1: Safety Lead-In (Cetuximab, Cis or Carbo, 5-FU): Combination Therapy (maximum 6 cycles):
  * United States (US) commercial cetuximab, manufactured by ImClone, 400 milligrams per square meter (mg/m^2) intravenous (IV) infusion on Day 1 of Cycle 1; subsequently 250 mg/m^2 IV infusion weekly.
  * Cisplatin (cis) 100 mg/m^2 or carboplatin (carbo) area under the curve (AUC) 5, up to a maximum 750 mg dose, IV infusion on Day 1 of every 21-day cycle, 1 hour after cetuximab infusion.
  * 5-Fluorouracil (5-FU): 1000 mg/m^2 IV infusion on Days 1 through 4 of every 21-day cycle.
  Monotherapy Therapy:
  Participants who did not experience disease progression after 6 cycles of combination therapy continued on weekly US commercial cetuximab monotherapy 250 mg/m^2 until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- Part 2: Cetuximab (US Commercial), Cis or Carbo, 5-FU: Combination Therapy (maximum 6 cycles):
  * US commercial cetuximab, manufactured by ImClone, 400 mg/m^2 IV infusion on Day 1 of Cycle 1; subsequently 250 mg/m^2 IV infusion weekly.
  * Cis 100 mg/m^2 or carbo AUC 5, up to a maximum 750 mg dose, IV infusion on Day 1 of every 21-day cycle, 1 hour after cetuximab infusion.
  * 5-FU: 1000 mg/m^2 IV infusion on Days 1 through 4 of every 21-day cycle.
  Monotherapy Therapy:
  Participants who did not experience disease progression after 6 cycles of combination therapy continued on weekly US commercial cetuximab monotherapy 250 mg/m^2 until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- Part 2: Cetuximab (Manufactured by BI), Cis or Carbo, 5-FU: Combination Therapy (maximum 6 cycles):
  * Cetuximab, manufactured by Boehringer Ingelheim (BI), 400 mg/m^2 IV infusion on Day 1 of Cycle 1; subsequently 250 mg/m^2 IV infusion weekly.
  * Cis 100 mg/m^2 or carbo AUC 5, up to a maximum 750 mg dose, IV infusion on Day 1 of every 21-day cycle, 1 hour after cetuximab infusion.
  * 5-FU: 1000 mg/m^2 IV infusion on Days 1 through 4 of every 21-day cycle.
  Monotherapy Therapy:
  Participants who did not experience disease progression after 6 cycles of combination therapy continued on weekly BI-manufactured cetuximab monotherapy 250 mg/m^2 until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
Period: Overall Study
Arm/Group | Part 1: Safety Lead-In (Cetuximab, Cis or Carbo, 5-FU) | Part 2: Cetuximab (US Commercial), Cis or Carbo, 5-FU | Part 2: Cetuximab (Manufactured by BI), Cis or Carbo, 5-FU
Started | 33 | 81 | 73
Received at Least 1 Dose of Study Drug | 33 | 77 | 71
Completed | 33 | 77 | 71
Not Completed | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of any study drug (cetuximab, cisplatin, carboplatin, or 5-FU).
Groups:
- Part 1: Safety Lead-In (Cetuximab, Cis or Carbo, 5-FU); Part 2: Cetuximab (US Commercial), Cis or Carbo, 5-FU: Combination Therapy (maximum 6 cycles):
  * US commercial cetuximab, manufactured by ImClone, 400 mg/m^2 IV infusion on Day 1 of Cycle 1; subsequently 250 mg/m^2 IV infusion weekly.
  * Cis 100 mg/m^2 or carbo AUC 5, up to a maximum 750 mg dose, IV infusion on Day 1 of every 21-day cycle, 1 hour after cetuximab infusion.
  * 5-FU: 1000 mg/m^2 IV infusion on Days 1 through 4 of every 21-day cycle.
  Monotherapy Therapy:
  Participants who did not experience disease progression after 6 cycles of combination therapy continued on weekly US commercial cetuximab monotherapy 250 mg/m^2 until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- Part 2: Cetuximab (Manufactured by BI), Cis or Carbo, 5-FU: Combination Therapy (maximum 6 cycles):
  * Cetuximab, manufactured by BI, 400 mg/m^2 IV infusion on Day 1 of Cycle 1; subsequently 250 mg/m^2 IV infusion weekly.
  * Cis 100 mg/m^2 or carbo AUC 5, up to a maximum 750 mg dose, IV infusion on Day 1 of every 21-day cycle, 1 hour after cetuximab infusion.
  * 5-FU: 1000 mg/m^2 IV infusion on Days 1 through 4 of every 21-day cycle.
  Monotherapy Therapy:
  Participants who did not experience disease progression after 6 cycles of combination therapy continued on weekly BI-manufactured cetuximab monotherapy 250 mg/m^2 until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- Total: Total of all reporting groups
Arm/Group | Part 1: Safety Lead-In (Cetuximab, Cis or Carbo, 5-FU) | Part 2: Cetuximab (US Commercial), Cis or Carbo, 5-FU | Part 2: Cetuximab (Manufactured by BI), Cis or Carbo, 5-FU | Total
Number analyzed (Participants) | 33 | 77 | 71 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (8.74) | 57.1 (10.75) | 59.4 (10.49) | 59.0 (10.47)
Sex/Gender, Customized [Number; unit: participants]
  Female | 11 | 9 | 15 | 35
  Male | 22 | 68 | 55 | 145
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 16 | 9 | 27
  Asian | 0 | 1 | 2 | 3
  Black or African American | 2 | 7 | 2 | 11
  White | 29 | 53 | 56 | 138
  More than 1 race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants] — Region of enrollment not available for 1 participant in the cetuximab manufactured by BI reporting group; N=70.
  participants
    United States | 27 | 25 | 28 | 80
    Mexico | 1 | 23 | 15 | 39
    Canada | 5 | 29 | 27 | 61
Disease Stage at Study Entry [Number; unit: participants]
  Locoregional | 6 | 34 | 32 | 72
  Metastatic | 27 | 43 | 38 | 108
  Unknown or not reported | 0 | 0 | 1 | 1
Karnofsky Performance Status (KPS) [Number; unit: participants] — The KPS rates the performance status and neurological functioning of a participant on a scale from KPS 0 (Dead) to KPS 100 (No complaints; no evidence of disease) in increments of 10. KPS 90 (Able to carry on normal activity; minor signs or symptoms of disease), KPS 80 (Normal activity with effort; some signs or symptoms of disease), and KPS 70 (Cares for self; unable to carry on normal activity or do active work).
  participants
    KPS 70 | 5 | 9 | 7 | 21
    KPS 80 | 19 | 28 | 22 | 69
    KPS 90 | 5 | 32 | 31 | 68
    KPS 100 | 4 | 8 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Treatment-Emergent Adverse Events (TEAEs); Data Analysis Cut-Off: September 27, 2013
Description: September 27, 2013 is the date when data was last collected for the primary endpoint. Prior to this date, the manufacturing process for the BI-manufactured cetuximab was changed necessitating the need to switch participants to US commercial cetuximab. All other components of their treatment regimen remained unchanged and participants stayed in their original reporting group. Therefore, the number of participants in the BI-manufactured cetuximab treatment arm who had TEAEs includes TEAEs while participants received BI-manufactured and US-commercial cetuximab. Using September 27 cut-off, the analysis of TEAEs is confounded by the switch from BI-manufactured to US commercial cetuximab. TEAEs were defined as serious and other non-serious AEs that occurred or worsened after study treatment (regardless of causality). TEAE information for Safety Lead-In group available in Reported Adverse Events module which is summary of serious and other non-serious AEs regardless of causality.
Time Frame: Part 2: Baseline to end of combination therapy (up to 18 weeks)
Population: Participants who received at least 1 dose of study drug (cetuximab, cisplatin, carboplatin, or 5-FU) according to the treatment arm to which they were assigned or randomized. Data is confounded for 9 participants in BI-manufactured cetuximab treatment arm who switched to US commercial cetuximab.
Measure: Number; unit: participants
Groups:
- Part 2: Combination Therapy: Cetuximab (US Commercial): Combination Therapy (maximum 6 cycles):
  * US commercial cetuximab, manufactured by ImClone, 400 mg/m^2 IV infusion on Day 1 of Cycle 1; subsequently 250 mg/m^2 IV infusion weekly.
  * Cis 100 mg/m^2 or carbo AUC 5, up to a maximum 750 mg dose, IV infusion on Day 1 of every 21-day cycle, 1 hour after cetuximab infusion.
  * 5-FU: 1000 mg/m^2 IV infusion on Days 1 through 4 of every 21-day cycle.
- Part 2: Combination Therapy: Cetuximab (Manufactured by BI): Combination Therapy (maximum 6 cycles):
  * Cetuximab, manufactured by BI, 400 mg/m^2 IV infusion on Day 1 of Cycle 1; subsequently 250 mg/m^2 IV infusion weekly.
  * Cis 100 mg/m^2 or carbo AUC 5, up to a maximum 750 mg dose, IV infusion on Day 1 of every 21-day cycle, 1 hour after cetuximab infusion.
  * 5-FU: 1000 mg/m^2 IV infusion on Days 1 through 4 of every 21-day cycle.
Arm/Group | Part 2: Combination Therapy: Cetuximab (US Commercial) | Part 2: Combination Therapy: Cetuximab (Manufactured by BI)
Number analyzed (Participants) | 77 | 71
participants | 76 | 68

2. Primary Outcome: Number of Participants Who Had TEAEs; Data Analysis Cut-Off: January 23, 2013
Description: January 23, 2013 is the date when the first participant in the BI-manufactured cetuximab treatment arm switched to US commercial cetuximab due to changes in the manufacturing process for the BI-manufactured cetuximab necessitating the need to switch participants to US commercial cetuximab. Each participant who switched treatments received at least 2 cycles of BI-manufactured cetuximab before switching. All other components of their treatment regimen remained unchanged. The number of participants who had TEAEs during combination therapy is reported. Using January 23 cut-off, data is un-confounded by lack of BI-manufactured cetuximab. TEAEs were defined as serious and other non-serious adverse events (AEs) that occurred or worsened after study treatment (regardless of causality). TEAE information for Safety Lead-in group available in Reported Adverse Event module which is summary of serious and other non-serious AEs regardless of causality.
Time Frame: Part 2: Baseline to end of combination therapy or date first participant switched to US commercial cetuximab (up to 18 weeks)
Population: Participants who received at least 1 dose of study drug (cetuximab, cisplatin, carboplatin, or 5-FU) according to the treatment arm to which they were assigned or randomized.
Measure: Number; unit: participants
Groups:
- Part 2: Combination Therapy: Cetuximab (Manufactured by BI),: Combination Therapy (maximum 6 cycles):
  * Cetuximab, manufactured by BI, 400 mg/m^2 IV infusion on Day 1 of Cycle 1; subsequently 250 mg/m^2 IV infusion weekly.
  * Cis 100 mg/m^2 or carbo AUC 5, up to a maximum 750 mg dose, IV infusion on Day 1 of every 21-day cycle, 1 hour after cetuximab infusion.
  * 5-FU: 1000 mg/m^2 IV infusion on Days 1 through 4 of every 21-day cycle.
Arm/Group | Part 2: Combination Therapy: Cetuximab (US Commercial) | Part 2: Combination Therapy: Cetuximab (Manufactured by BI),
Number analyzed (Participants) | 77 | 71
participants | 75 | 68

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as duration from the date of randomization to the date of death from any cause. For each participant not known to have died as of the 23 October 2014 data cutoff date for the analysis, OS was censored at the date last known to be alive. In addition, any participants on Arm B who was switched from BI-manufactured cetuximab to ImClone-manufactured cetuximab was censored at the time of the switch.
Time Frame: Parts 1 and 2: Randomization to Date of Death from any Cause (Up to 36.3 Months)
Population: All participants who received at least on dose of study drug. 4 participants were censored in Safety Lead-In, 17 participants were censored in Cetuximab (US Commercial) and 15 in Cetuximab (Manufactured by BI).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Part 2: Combination Therapy: Cetuximab (Manufactured by BI): Combination Therapy (maximum 6 cycles):
  * Cetuximab, manufactured by Boehringer Ingelheim (BI), 400 mg/m^2 IV infusion on Day 1 of Cycle 1; subsequently 250 mg/m^2 IV infusion weekly.
  * Cis 100 mg/m^2 or carbo AUC 5, up to a maximum 750 mg dose, IV infusion on Day 1 of every 21-day cycle, 1 hour after cetuximab infusion.
  * 5-FU: 1000 mg/m^2 IV infusion on Days 1 through 4 of every 21-day cycle.
Arm/Group | Part 1: Safety Lead-In (Cetuximab, Cis or Carbo, 5-FU) | Part 2: Combination Therapy: Cetuximab (US Commercial) | Part 2: Combination Therapy: Cetuximab (Manufactured by BI)
Number analyzed (Participants) | 33 | 77 | 71
Months | 9.13 [6.60 to 10.38] | 9.23 [6.90 to 11.80] | 9.46 [6.87 to 11.43]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as duration from the date of randomization to the first date of objective progressive disease (PD) or death from any cause. For each participant who was not known to have died or to have had objective PD as of the 23 October 2014 data cutoff date for the analysis, PFS was censored at the date of the participant's last complete tumor assessment prior to that cutoff date. In addition, any participant in Arm B who was switched from BI-manufactured cetuximab to ImClone-manufactured cetuximab was censored at the time of the switch.
Time Frame: Parts 1 and 2: Randomization to Progression of Disease or Death from any Cause (Up to 32.7 Months)
Population: All participants who received at least one dose of study drug. 7 participants were censored in Safety Lead-In ,12 participants were censored in Cetuximab (US Commercial) and 15 in Cetuximab (Manufactured by BI).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: Safety Lead-In (Cetuximab, Cis or Carbo, 5-FU) | Part 2: Combination Therapy: Cetuximab (US Commercial) | Part 2: Combination Therapy: Cetuximab (Manufactured by BI)
Number analyzed (Participants) | 33 | 77 | 71
Months | 4.57 [3.22 to 5.32] | 4.34 [3.52 to 5.78] | 5.59 [4.04 to 6.28]

5. Secondary Outcome: Percentage of Participants Having a Confirmed Best Response of Complete Response (CR) or Partial Response (PR) (Overall Response Rate [ORR])
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version [v]1.0) criteria. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions. Percentage of participants with a confirmed CR or PR=(number of participants whose best overall response was CR or PR)/(number of participants treated)*100.
Time Frame: Parts 1 and 2: Randomization to Progression of Disease (Up to 32.7 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Safety Lead-In (Cetuximab, Cis or Carbo, 5-FU) | Part 2: Combination Therapy: Cetuximab (US Commercial) | Part 2: Combination Therapy: Cetuximab (Manufactured by BI)
Number analyzed (Participants) | 33 | 77 | 71
percentage of participants | 24.2 [9.6 to 38.9] | 32.5 [22.0 to 42.9] | 36.6 [25.4 to 47.8]

6. Secondary Outcome: Number of Participants With Anti-Cetuximab Antibodies
Time Frame: Day 1, Week 1 of Cycles 3 and 5 (postbaseline samples were collected prior to infusion).
Population: Participants who received at least 1 dose of study drug and had evaluable data for antibodies.There was no pre-specified analysis plan for trial to report immunogenicity results separately for each arm,as results were intended to be pooled and combined with other cetuximab trials data.Data was pooled for the three arms for cetuximab in this trial.
Measure: Number; unit: participants
Groups:
- All Participants (Cetuximab): United States (US) commercial cetuximab, manufactured by ImClone, 400 milligrams per square meter (mg/m^2) intravenous (IV) infusion on Day 1 of Cycle 1; subsequently 250 mg/m^2 IV infusion weekly.
  OR
  Cetuximab, manufactured by Boehringer Ingelheim (BI), 400 mg/m^2 IV infusion on Day 1 of Cycle 1; subsequently 250 mg/m^2 IV infusion weekly.
Arm/Group | All Participants (Cetuximab)
Number analyzed (Participants) | 85
participants | 4

7. Secondary Outcome: Percentage of Participants Having a Best Response of CR, PR, or Stable Disease (SD) - Disease Control Rate (DCR)
Description: Response was defined using RECIST, v1.0 criteria. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions. Progressive Disease (PD) was defined as having at least a 20% increase in the sum of the longest diameter of target lesions. Stable Disease (SD) was defined as small changes that did not meet the above criteria.
Time Frame: Parts 1 and 2: Randomization to Progression of Disease (Up to 32.7 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Safety Lead-In (Cetuximab, Cis or Carbo, 5-FU) | Part 2: Combination Therapy: Cetuximab (US Commercial) | Part 2: Combination Therapy: Cetuximab (Manufactured by BI)
Number analyzed (Participants) | 33 | 77 | 71
percentage of participants | 69.7 [54.0 to 85.4] | 58.4 [47.4 to 69.4] | 62.0 [50.7 to 73.3]

8. Secondary Outcome: Maximum Serum Concentration (Cmax) of Cetuximab Following 400 mg/m² Cetuximab Dosing
Description: The Cmax of cetuximab following 400 mg/m² cetuximab dosing during Part 2 of the study is reported. As specified in the protocol, pharmacokinetics (PK) samples were not collected during Part 1 of the study, Safety Lead-In or during Part 2 monotherapy.
Time Frame: Part 2: Cycle 1, Day 1: 0 hours [(h); immediately postdose], 1 h, 2 h, and 24 h postdose
Population: Participants who received at least 1 dose of cetuximab (400 mg/m²) and had valid serum cetuximab concentrations during the specified time frame. No participant was analyzed during Part 1 of the study, Safety Lead-In or during Part 2 monotherapy..
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Part 2: Combination Therapy: Cetuximab (US Commercial) | Part 2: Combination Therapy: Cetuximab (Manufactured by BI)
Number analyzed (Participants) | 61 | 53
micrograms per milliliter (μg/mL) | 208 (10.2) | 208 (7.8)

9. Secondary Outcome: Cmax of Cetuximab at Steady State
Description: A total of 4 samples were collected at various times during combination therapy, from the third dose of 250 mg/m^2 cetuximab in Cycle 1 (Week 3) through the final dose in Cycle 3 (Week 3) and used to report Cmax of cetuximab at steady state during Part 2 of the study. As specified in the protocol, PK samples were not collected during Part 1 of the study, Safety Lead-In, or during Part 2 monotherapy.
Time Frame: Part 2: Weekly from Cycle 1, Week 3 through Cycle 3, Week 3: 0 h (immediately postdose), 24 h, 96 h, and 168 h postdose
Population: Participants who received at least 1 dose of cetuximab (400 mg/m^2) and had valid serum cetuximab concentrations during the specified time frame. No participant was analyzed during Part 1 of the study, Safety Lead-In, or during Part 2 monotherapy.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Part 2: Combination Therapy: Cetuximab (US Commercial) | Part 2: Combination Therapy: Cetuximab (Manufactured by BI)
Number analyzed (Participants) | 44 | 46
micrograms per milliliter (μg/mL) | 225 (17.7) | 199 (15.3)

10. Secondary Outcome: Area Under the Concentration Curve (AUC) of Cetuximab at Steady State
Description: A total of 4 samples were collected during combination therapy, from the first dose of 250 mg/m^2 cetuximab in Cycle 1 (Day 1) through the final dose in Cycle 3 (Week 3) and used to report AUC of cetuximab at steady state during Part 2 of the study. As specified in the protocol, PK samples were not collected during Part 1 of the study, Safety Lead-In, or during Part 2 monotherapy.
Time Frame: Part 2: Weekly from Cycle 1, Day 1 through Cycle 3, Week 3: 0 h (immediately postdose), 24 h, 96 h, and 168 h postdose
Population: Participants who received at least 1 dose of cetuximab (250 mg/m^2) and had valid serum cetuximab concentrations during the specified time frame. No participant was analyzed during Part 1 of the study, Safety Lead-In, or during Part 2 monotherapy.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours/milliliter (μg*h/mL)
Arm/Group | Part 2: Combination Therapy: Cetuximab (US Commercial) | Part 2: Combination Therapy: Cetuximab (Manufactured by BI)
Number analyzed (Participants) | 61 | 55
micrograms*hours/milliliter (μg*h/mL) | 21900 (31.8) | 18800 (25.5)

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and other non-serious AEs are reported for participants who received at least 1 dose of any drug (cetuximab, cisplatin, carboplatin, or 5-FU). Death due to progressive disease was not considered an AE.
Arm/Group | Part 1: Safety Lead-In (Cetuximab, Cis or Carbo, 5-FU) | Part 2: Cetuximab (US Commercial), Cis or Carbo, 5-FU | Part 2: Cetuximab (Manufactured by BI), Cis or Carbo, 5-FU
Serious Adverse Events (participants affected / at risk) | 20/33 | 48/77 | 42/71
Other Adverse Events (participants affected / at risk) | 32/33 | 64/77 | 62/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Safety Lead-In (Cetuximab, Cis or Carbo, 5-FU) (N=33) | Part 2: Cetuximab (US Commercial), Cis or Carbo, 5-FU (N=77) | Part 2: Cetuximab (Manufactured by BI), Cis or Carbo, 5-FU (N=71)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 4 (8) | 5 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (2) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (5) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 6 (9) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (3) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 3 (5) | 2 (5)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (10) | 2 (2)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (4) | 7 (10) | 4 (7)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (10) | 1 (1) | 1 (2)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 4 (5) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1)
Thrombosis in device (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (3) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 3 (3) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (3)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Device related infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (4)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Joint abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (6) | 5 (9) | 5 (6)
Sepsis (Infections and infestations) | 3 (3) | 5 (5) | 1 (2)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 4 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (4) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Vena cava injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (4) | 1 (3) | 1 (1)
Platelet count decreased (Investigations) | 2 (3) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 1 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (8) | 7 (10) | 9 (11)
Fluid intake reduced (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (6) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6) | 3 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (4) | 0 (0)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (30)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 3 (5) | 2 (4)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 3 (9)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (5) | 1 (3)
Embolism (Vascular disorders) | 2 (3) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (8) | 0 (0) | 2 (3)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part 1: Safety Lead-In (Cetuximab, Cis or Carbo, 5-FU) (N=33) | Part 2: Cetuximab (US Commercial), Cis or Carbo, 5-FU (N=77) | Part 2: Cetuximab (Manufactured by BI), Cis or Carbo, 5-FU (N=71)
Anaemia (Blood and lymphatic system disorders) | 18 (86) | 19 (103) | 27 (138)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (17)
Leukopenia (Blood and lymphatic system disorders) | 3 (8) | 4 (19) | 4 (13)
Neutropenia (Blood and lymphatic system disorders) | 15 (60) | 17 (30) | 23 (64)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (35) | 6 (8) | 10 (39)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 5 (18)
Ear pain (Ear and labyrinth disorders) | 3 (14) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 6 (68) | 8 (62)
Eye pruritus (Eye disorders) | 3 (8) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 4 (13)
Abdominal pain (Gastrointestinal disorders) | 4 (12) | 6 (18) | 6 (19)
Constipation (Gastrointestinal disorders) | 9 (31) | 16 (48) | 25 (112)
Diarrhoea (Gastrointestinal disorders) | 15 (39) | 23 (47) | 22 (49)
Dry mouth (Gastrointestinal disorders) | 2 (15) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (28) | 8 (25)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (24)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (28) | 7 (32) | 7 (57)
Glossodynia (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 19 (88) | 34 (109) | 33 (102)
Oral pain (Gastrointestinal disorders) | 0 (0) | 5 (21) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 9 (36) | 21 (96) | 22 (114)
Vomiting (Gastrointestinal disorders) | 15 (35) | 17 (44) | 25 (82)
Asthenia (General disorders) | 2 (3) | 8 (49) | 4 (15)
Chest pain (General disorders) | 2 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 16 (91) | 35 (204) | 37 (221)
Mucosal inflammation (General disorders) | 5 (24) | 12 (41) | 16 (83)
Oedema peripheral (General disorders) | 3 (5) | 0 (0) | 5 (18)
Pain (General disorders) | 0 (0) | 5 (14) | 4 (12)
Pyrexia (General disorders) | 5 (9) | 8 (10) | 8 (9)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (10)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (8) | 0 (0)
Paronychia (Infections and infestations) | 2 (5) | 9 (74) | 10 (63)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (14)
Upper respiratory tract infection (Infections and infestations) | 2 (9) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (6) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1/11 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 3 (14) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 7 (9) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 2 (4) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (15) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (22) | 11 (26) | 14 (35)
Platelet count decreased (Investigations) | 5 (14) | 11 (51) | 10 (48)
Weight decreased (Investigations) | 7 (34) | 10 (58) | 14 (65)
White blood cell count decreased (Investigations) | 6 (15) | 0 (0) | 4 (9)
Decreased appetite (Metabolism and nutrition disorders) | 6 (26) | 15 (70) | 21 (69)
Dehydration (Metabolism and nutrition disorders) | 8 (17) | 8 (12) | 12 (23)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (23) | 4 (9) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (24) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (17) | 4 (25) | 7 (22)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (31) | 17 (69) | 23 (82)
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 (73) | 30 (237) | 29 (161)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (10) | 0 (0) | 10 (38)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 4 (11) | 8 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (31) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (13) | 5 (9) | 4 (12)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 9 (41)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (13) | 5 (25)
Dizziness (Nervous system disorders) | 3 (16) | 9 (43) | 11 (29)
Dysgeusia (Nervous system disorders) | 6 (30) | 4 (12) | 8 (27)
Headache (Nervous system disorders) | 2 (5) | 7 (37) | 6 (10)
Neuropathy peripheral (Nervous system disorders) | 2 (9) | 0 (0) | 6 (19)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (21) | 0 (0) | 7 (55)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 5 (6)
Anxiety (Psychiatric disorders) | 2 (6) | 0 (0) | 5 (17)
Confusional state (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 4 (29) | 6 (24)
Insomnia (Psychiatric disorders) | 3 (28) | 10 (78) | 11 (80)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 4 (22) | 9 (39)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (14) | 10 (90) | 13 (80)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 6 (43) | 6 (21)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (10) | 5 (16) | 5 (14)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (17) | 7 (44)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 17 (101) | 26 (254) | 19 (134)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (17) | 19 (142) | 12 (87)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (9) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (11) | 8 (60) | 6 (27)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (17) | 4 (34) | 5 (22)
Rash (Skin and subcutaneous tissue disorders) | 7 (41) | 11 (91) | 19 (152)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (13) | 5 (31)
Skin fissures (Skin and subcutaneous tissue disorders) | 3 (8) | 6 (48) | 8 (48)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (6) | 4 (9) | 5 (14)
Embolism (Vascular disorders) | 0 (0) | 4 (37) | 0 (0)
Hypertension (Vascular disorders) | 2 (26) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (9) | 10 (27) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days